CLINICAL TRIAL: NCT02904694
Title: Commissioning Through Evaluation: Selective Dorsal Rhizotomy Database
Brief Title: Selective Dorsal Rhizotomy (SDR) Database
Acronym: SDR
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 162253
Record Dates: First submitted 2016-07-14; First posted 2016-09-19 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2017-12

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A national database is being set-up to collate clinical outcome information before and after children undergo Selective Dorsal Rhizotomy (SDR). SDR is a surgical procedure that has been used for many years but has not been routinely available within the United Kingdom National Health Service (NHS). The SDR procedure is used to improve spasticity in children with cerebral palsy and involves dividing some of the nerve fibres running from the muscles back to the spinal cord. While it is believed that SDR is effective, there are no definitive data. In July 2014 NHS England commissioned five NHS Trusts to undertake SDR surgery in eligible children for a two-year period, and to collect detailed information on their outcomes. The proposed database will aggregate these data from the five centres and analyse them to provide overall evidence on the clinical effectiveness of SDR. This information will be used to inform future commissioning decisions. The database has been developed by the King's Technology Evaluation Centre (KiTEC) in conjunction with NHS England and the national clinical SDR steering committee and its data subcommittee. KiTEC undertakes research evaluations for the National Institute for Health and Care Excellence (NICE), and has been commissioned by NICE to undertake this work. Clinicians in the SDR data subgroup have liaised closely with KiTEC to agree which data to collect so that it the least amount needed and will be in a standardised format across all centres. When all two-year outcome data are recorded, KiTEC will analyse the data and present a report to NHS England, NICE and the SDR steering committee and data sub-group. While there are no firm plans to follow the children beyond two years post-surgery, all parties involved are hoping that further funding can be obtained to continue following these children up as these data will be unique.

DETAILED DESCRIPTION:
Disease overview:

Cerebral Palsy is an all-encompassing term for numerous neurological conditions caused by problems in the brain and nervous system. More specifically, cerebral palsy is related to problems in muscle movement, which result in abnormalities in walking, posture, and balance. Other important functions can also be affected, such as language/communication, learning, and vision. There is currently no cure for cerebral palsy; however, there are several treatment options that can aid alleviation of symptoms and improve quality of life. The selection of appropriate treatment(s) for each child requires input from a multi-disciplinary team of health professionals, such as paediatricians, social workers, physiotherapists, speech and language therapists, occupational therapists, neurologists and surgeons.

Treatment overview:

The National Institute for Health and Care Excellence (NICE) published guidance related to treatment options for cerebral palsy in 2012 (CG145). One of the treatment options discussed was Selective Dorsal Rhizotomy (SDR). SDR is an irreversible surgical procedure, which involves the division of some of the sensory nerves of the spinal cord in order to reduce sensory input to the sensory-motor reflex arcs. Intensive physiotherapy is required SDR post surgery for up to 24 months to achieve the outcome goals of improvement in muscle function, tone, and quality of life. NICE CG145 recommends consideration of SDR in children with a GMFCS level II or III. This recommendation was based on a review of evidence evaluation, which concluded that there was reasonable evidence that SDR combined with appropriate post-operative treatment can result in significant improvements in motor function and quality of life.

Study Overview:

This current project is being commissioned by NICE to support NHS England in its Commissioning through Evaluation (CTE) approach. CTE was launched in September 2013 and involves funding medical treatments and technologies not routinely commissioned within the NHS. SDR is one such procedure which was selected for CTE, with the aim of evaluating the 'outcome of SDR and demonstrate improvement in function after SDR at 6 months that is maintained or improved at 12 months and two years post operation'. As part of this programme, NICE commissioned, in early 2014, a data collection and register development service from one of its External Assessment Centres (EACs): King's Imaging Technology Evaluation Centre (KiTEC). The key objective of the KiTEC EAC is to collect SDR related data that will inform clinical effectiveness and other outcomes of interest to NHS England in making its commissioning plans and addressing the following research question from section 4.5 of CG145:

'Does selective dorsal rhizotomy followed by intensive rehabilitation performed between the ages of 3 and 9 years in children who are at GMFCS level II or III result in good community mobility as a young adult?'

Study Design:

This is a multi-centre national database (register) project to obtain the evidence related to SDR that will address the research question in section 4.5 of CG145 and inform clinical effectiveness and other outcomes of interest to NHS England. All patients will undergo pre-assessment prior to undergoing SDR. This varies between centres, and can be anywhere from 6 months prior to SDR. Hospital admission for SDR usually is between 1-2 weeks. Post-SDR follow-up will be conducted up to two years for the purposes of this project. All patients' will followed up to two years post-SDR by members of the relevant clinical team. Post-SDR discharge there will be three main data collection points for the purposes of this project: 6, 12 and 24 months post-SDR. Patient data will be collected at various time-points, as agreed between the EAC and various SDR subgroup members. Pre-assessments may be split into more than one appointment, depending on the particular patient care pathway at each participating centre.

Parents of patients will be approached by the SDR clinical team when they attend for their first pre-SDR clinic visit. It will be explained to the parents and children that their hospital will be making clinical assessments before and after SDR to enable them to provide optimum care and to evaluate the success of the operation and post-operative rehabilitation. These assessments along with patient-reported outcomes, such as quality of life assessments, will be standardised across all five commissioned hospitals. The parents and children will be asked for permission to add their data to the national database to facilitate aggregation of results across the United Kingdom (UK).

Study information sheets will be provided. If they agree to take part, parents will sign a consent form at the 2nd pre-SDR visit. This will allow time for them to consider whether or not they wish to take part.

Centre and Subject Compliance:

Centre compliance refers to all centres providing the agreed standardised dataset and input into the standardised database as per the CTE selection criteria. The EAC will regularly monitor Centre compliance in liaison with NHS England and include tables of compliance in the project report. The project report (with potential for interim analysis) will include tables on the number of eligible patients that were referred for treatment through the multi-disciplinary team process and consented to part of the database as well as those that were actually registered in the SDR database. The project report (with potential for interim analysis) will list the percentage of missing data in each of the clinical domains and differentiate between baseline and follow-up variables. Depending on the stage of the database a table depicting the number of children that have been lost to follow up will be included in the project report or in potential interim analyses reports. The SDR centres will be given regular reports on the quality of their data in terms of missing variables and possible outliers.

Statistical Considerations:

The EAC statisticians will carry out all analyses. All data obtained will be analysed at regular specified time points to inform ongoing assessment of the clinical effectiveness, relevant outcomes and assessment of the overall research question.The SDR database is expected to have small numbers, in the region of up to n=120 a year in England. A range of clinical and patient-reported outcomes will be recorded and there will be no single primary or secondary outcome. Rather the aim is to describe and quantify the changes in a number of important clinical domains such as spasticity, function, range of motion, gait and quality of life.

Ethical Considerations:

As the database constitutes research involving human subjects, the following ethical considerations arise:

* Parental consent will be required to add the child's data to the national database and patient information sheets (PIS) have been developed for both children and parents of potential children at the designated SDR centres.
* Only the minimum number of data items needed to meet the objectives of the database and comply with ethical and regulatory requirements will be included in the final dataset.
* Children's confidentiality will be protected during data collection and handling thus reducing the risk of disclosure.

ELIGIBILITY:
Inclusion Criteria:

All patients who have consented to the SDR procedure in one of the five Trusts who are commissioned to do SDR.

These will be asked to consent to their outcome data being added to the national database. There are no exclusions to the database.

For inclusion in the CTE SDR programme, the criteria were established as:

* Children between the ages of 3 and 9 years with a diagnosis of spastic diplegic cerebral palsy (based on NICE guidance [2]).
* Dynamic spasticity in lower limbs affecting function and mobility and no dystonia
* MRI shows typical Cerebral palsy changes and no damage to key areas of brain controlling posture and coordination.
* GMFCS level II or III.
* No evidence of genetic or neurological progressive illness.
* Mild to moderate lower limb weakness with ability to maintain antigravity postures.
* No significant scoliosis or hip dislocation (Reimer's index [10] should be <40%).
* In addition to the above clinical criteria there must be written agreement from the referring responsible commissioner confirming financial and resource commitment to provide the post operative physiotherapy package as outlined in the CTE SDR programme selection criteria [5].

Exclusion Criteria:

* Under 3 years of age, or older than 9 years.
* Gross Motor Function Classification System levels I, IV or V.
* Any other medical or personal aspects in conflict with those listed above under inclusion criteria.

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients who have consented to the Selective Dorsal Rhizotomy (SDR) procedure in one of the five Trusts who are commissioned to do SDR.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2014-03; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Change in Gross Motor Function Measure (GMFM-66) | Change from baseline, to 6 months, 12 months and 24 months.
  The GMFM-66 is a clinical tool to evaluate gross mortar function change in children with cerebral palsy. It contains 66 items in the tool, which a aggregated using a predefined summary calculation of all completed items.
Change in the Cerebral Palsy Quality of Life Questionnaire for Children | Change from Baseline, to 6 months, 12 months and 24 months
  The Change in the Cerebral Palsy Quality of Life Questionnaire for Children, is a quality of life measure for children with cerebral palsy which can be completed by either the child, or the parent. It contains 53 items in the child version, and 65 items in the parent version.

SECONDARY OUTCOMES:
Duncan Ely Test: used to assess rectus femoris spasticity or tightness | Change from Baseline, to 6 months, 12 months and 24 months
Modified Ashworth Scale | Change from Baseline, to 6 months, 12 months and 24 months
Physiotherapy assessment measures: use of mobility and orthotic devices, and functional mobility scale. | Change from Baseline, to 6 months, 12 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Janet Peacock, PhD, Principal Investigator — King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided